CLINICAL TRIAL: NCT03622658
Title: A Phase 2a Study to Evaluate the Safety and Efficacy of Namilumab in Subjects With Moderate-to-severely Active Axial Spondyloarthritis
Brief Title: Efficacy and Safety of Namilumab for Moderate-to-severe Axial Spondyloarthritis
Acronym: NAMASTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Izana Bioscience Ltd. (Industry)
Collaborators: Iqvia Pty Ltd (Industry); Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IZN-101
Record Dates: First submitted 2018-07-17; First posted 2018-08-09 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-01

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — namilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo solution administered by subcutaneous injection on 4 occasions over 10 weeks
  Interventions: Biological: Placebo
- Namilumab (Experimental): Namilumab (150 mg) administered by subcutaneous injection on 4 occasions over 10 weeks
  Interventions: Biological: Namilumab

INTERVENTIONS:
Biological: Placebo — Placebo solution for subcutaneous injection.
  Arms: Placebo
Biological: Namilumab — Namilumab solution for subcutaneous injection
  Arms: Namilumab

SUMMARY:
The study will assess the effect of namilumab, a GM-CSF inhibitor, on the clinical response in subjects with axial spondyloarthritis. Subjects will receive treatment with either namilumab or placebo.

DETAILED DESCRIPTION:
A phase 2a proof-of-concept, randomised, double-blind, placebo-controlled study to evaluate the safety/tolerability and efficacy of 4 subcutaneous injections of namilumab (150 mg) given over 10 weeks in subjects with moderate-to-severely active axial spondyloarthritis including those previously exposed to anti- TNF therapy (NAMASTE study).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years of age.
* Diagnosis of axSpA by an appropriately qualified physician and classified using ASAS criteria ≥ 3 months prior to Baseline.
* Bath Ankylosing Spondylitis Disease Activity Index score ≥ 4 and spinal pain score ≥ 40, at screening and Baseline.
* MRI evidence of active axSpA ≤ 6 (ideally ≤ 3) months prior to randomisation using ASAS criteria.
* Stable NSAID use prior to study entry.
* Stable use of MTX, sulfasalazine or leflunomide prior to study entry.
* Stable oral corticosteroid dose prior to study entry.
* Capable of giving signed informed consent.
* Inadequately responded to or experienced intolerance to previous treatment with an anti-TNF agent (some subjects).

Exclusion Criteria:

* Current diagnosis of axSpA with a BASDAI > 4 but no evidence of inflammation on MRI.
* Discontinued biologic therapy < 8 weeks prior to Baseline.
* Previous or current use of oral corticosteroid as defined in protocol.
* Received intra-articular or i.v. corticosteroids prior to or during Screening.
* Received anti-IL-17A or anti-IL-12/23 therapy.
* Received cyclosporine, tacrolimus or mycophenolate mofetil prior to Baseline.
* Previously received stem cell transplantation.
* Infection(s) requiring treatment with i.v. anti-infectives or oral anti-infectives prior to Baseline.
* Abnormal screening laboratory and other analyses.
* Receipt of any live vaccine within 2 weeks prior to randomisation, or will require live vaccination during study participation.
* Evidence of current or prior dysplasia or history of malignancy.
* Has had any uncontrolled and/or clinically significant illness, hospitalisation, or any surgical procedure requiring general anaesthesia prior to Screening, or any planned surgical procedure within 6 months after randomisation.
* Known current or previous interstitial lung disease.
* Positive pregnancy test at Screening (serum) or Baseline (urine).
* Female subjects who are breastfeeding or considering becoming pregnant during the study.
* Considered by the Investigator to be an unsuitable candidate for the study.
* Received any investigational agent or procedure within 30 days or 5 half-lives prior to Baseline.
* Related to or a dependent of the site staff, or a member of the site staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Taylor, PhD, Principal Investigator — Botnar Research Centre, University of Oxford
Locations (9):
- United Kingdom (9):
  - Royal United Hospitals Bath, Bath
  - University Hospital Birmingham, Birmingham
  - University Hospital Coventry and Warwickshire, Coventry
  - Northwick Park Hospital, London
  - Whipps Cross Hospital, London
  - Norfolk and Norwich University Hospital, Norwich
  - Oxford University Hospital, Oxford
  - Royal Berkshire Hospital, Reading
  - Haywood Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Worth C, Al-Mossawi MH, Macdonald J, Fisher BA, Chan A, Sengupta R, Packham J, Gaffney K, Gullick N, Cook JA, Corn TH, Teh J, Machado PM, Taylor PC, Bowness P. Granulocyte-macrophage colony-stimulating factor neutralisation in patients with axial spondyloarthritis in the UK (NAMASTE): a randomised, double-blind, placebo-controlled, phase 2 trial. Lancet Rheumatol. 2024 Aug;6(8):e537-e545. doi: 10.1016/S2665-9913(24)00099-7. Epub 2024 Jun 25. PMID 38942047

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Namilumab
Started | 6 | 36
Completed | 3 | 32
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Namilumab | Total
Number analyzed (Participants) | 6 | 36 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 35 | 41
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 15 | 17
  Male | 4 | 21 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 33 | 38
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 34 | 39
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 6 | 36 | 42
Height [Median (Full Range); unit: cm] | 175.5 [159.2 to 180] | 173.5 [152 to 191.5] | 174.5 [152 to 191.5]
Weight [Median (Full Range); unit: kg] | 86.5 [53.2 to 98.8] | 80.5 [54.1 to 126] | 82.15 [53.2 to 126]
BMI [Median (Full Range); unit: kg/m^2] | 27.85 [18.2 to 33.5] | 27.6 [19.2 to 41.6] | 27.65 [18.2 to 41.6]
Prior use of anti-tumor necrosis factor (TNF) treatment [Number; unit: participants] | 1 | 6 | 7
Duration of disease <2years [Number; unit: participants] | 4 | 16 | 20

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Who Achieved ASAS20 Clinical Response
Description: The primary endpoint was the proportion of subjects who achieved an Assessment in Ankylosing Spondylitis with 20% improvement (ASAS20) clinical response at Week 12.
  An ASAS20 clinical response was defined as an improvement of at least 20% and an absolute improvement of at least 10 units on a 0 to 100 scale in at least three of the following four domains collected in the electronic case report form (eCRF) and no worsening in the fourth domain: Subject's Global Assessment of Disease Status, Subject's Assessment of Spinal Pain, function (Bath Ankylosing Spondylitis Functional Index [BASFI]) and inflammation (last two questions of the BASDAI). Lower values within the individual domains represent less severe symptoms.
Time Frame: Weeks 12
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Namilumab
Number analyzed (Participants) | 6 | 36
Participants | 3 | 14

2. Secondary Outcome: Proportion of Subjects Who Achieved ASAS40 Clinical Response at Week 12
Description: Proportion of subjects who achieved Assessment in Ankylosing Spondylitis with 40% improvement (ASAS40) response at Week 12
Time Frame: Week 12
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Namilumab
Number analyzed (Participants) | 6 | 36
Participants | 3 | 9

3. Secondary Outcome: Proportion of Subjects Who Achieved an ASAS20 Clinical Response at Week 6
Description: Proportion of subjects who achieved an ASAS20 clinical response at Week 6
Time Frame: Week 6
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Namilumab
Number analyzed (Participants) | 6 | 36
Participants | 0 | 12

4. Secondary Outcome: Proportion of Subjects Who Achieved Ankylosing Spondylitis Disease Activity Score C-reactive Protein (ASDAS-CRP) Response at Weeks 6
Description: Proportion (percentage) of subjects who achieved Ankylosing Spondylitis Disease Activity Score C-reactive Protein (ASDAS-CRP) response at Week 6, Clinically Important Improvement
Time Frame: Week 6
Population: Full Analysis Set. Overall number of participants analyzed reflect those with available ASDAS-CRP Scores as reported in the final clinical study report.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Namilumab
Number analyzed (Participants) | 5 | 33
Participants | 0 | 10

5. Secondary Outcome: Proportion of Subjects Who Achieved Clinically Important ASDAS-CRP Score at Week 12
Description: Proportion of Subjects Who Achieved Clinically Important ASDAS-CRP Score at Week 12, Clinically Important Improvement
Time Frame: Week 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Namilumab
Number analyzed (Participants) | 5 | 32
Participants | 1 | 10

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Placebo | Namilumab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/36
Other Adverse Events (participants affected / at risk) | 5/6 | 31/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Namilumab (N=36)
Duodenitis (Gastrointestinal disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=6) | Namilumab (N=36)
Macrocytosis (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 7
Frequent bowel movement (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Nasopharyngitis (Infections and infestations) | 0 | 9
Urinary tract infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Otitis externa (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3
Gastritis (Gastrointestinal disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypoaethesia (Nervous system disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Polymenorrhoea (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 2
Infected cyst (Infections and infestations) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Protein urine present (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03622658/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/58/NCT03622658/SAP_001.pdf